CLINICAL TRIAL: NCT06867952
Title: A Pilot Study of Vitamin K2 (Menaquinone-7, Soloways ™) in Patients With Osteopenia/Osteoporosis Carrying a VDR Gene Variant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW018
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteopenia; Osteoporosis; Supplements; Vitamin K2; Vitamin D
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Vitamin K 2; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): VDR Variant (Homozygous) Cohort
  Interventions: Dietary Supplement: Vitamin K2 plus vitamin D3
- Non-Variant (Control) Cohort (Experimental): Non-Variant (Control) Cohort
  Interventions: Dietary Supplement: Vitamin K2 plus vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin K2 plus vitamin D3 — Intervention: Vitamin K2 (menaquinone-7), 100-200 µg/day plus vitamin D3 (800- 1000 IU/day) for 6-9 months.
  Arms: Intervention
Dietary Supplement: Vitamin K2 plus vitamin D3 — Intervention: Vitamin K2 (menaquinone-7), 100-200 µg/day plus vitamin D3 (800- 1000 IU/day) for 6-9 months.
  Arms: Non-Variant (Control) Cohort

SUMMARY:
This pilot, genotype-stratified clinical trial aims to evaluate the safety and preliminary efficacy of vitamin K2 (menaquinone-7, MK-7) supplementation in patients with low bone mineral density (osteopenia or osteoporosis) who carry a specific "unfavorable" variant in the vitamin D receptor (VDR) gene (e.g., BsmI or ApaI polymorphisms). The trial will compare improvements in bone health and related biomarkers between two cohorts: (1) homozygous carriers of the VDR variant and (2) non-variant carriers (wild-type). Investigators hypothesize that MK-7 supplementation will lead to greater improvements in bone mineral density (BMD) and bone turnover markers in the homozygous variant group due to their potentially reduced baseline response to vitamin D signaling.

DETAILED DESCRIPTION:
Vitamin D receptor (VDR) polymorphisms have been associated with varying responses to vitamin D and calcium supplementation, ultimately influencing bone health. Menaquinone-7 (vitamin K2) is crucial for carboxylation of osteocalcin, facilitating calcium deposition in bone. This study investigates whether individuals with an "unfavorable" VDR gene variant - who might have lower basal responsiveness to vitamin D - experience enhanced benefit from MK-7 supplementation in conjunction with a standard vitamin D3 regimen. By focusing on this genotype-stratified approach, the study aims to generate preliminary data supporting the role of personalized supplementation strategies in skeletal health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-75 years with a confirmed DXA-based diagnosis of osteopenia or osteoporosis (T-score ≤ -1.0).
* Stable dietary habits and willingness to maintain current exercise regimen throughout the study.
* Willingness to undergo genotyping for the VDR variant. For the VDR Variant Cohort: confirmed homozygous "unfavorable" variant (e.g., BsmI or ApaI).
* For the Non-Variant Cohort: confirmed absence of the "unfavorable" allele (wild-type).

Exclusion Criteria:

* Current or recent (last 3 months) use of high-dose bisphosphonates, anabolic agents (e.g., teriparatide), or selective estrogen receptor modulators (SERMs). Known allergy or hypersensitivity to vitamin K or vitamin D supplements.
* Severe renal or hepatic dysfunction, uncontrolled hyperthyroidism, or other significant comorbidities that could confound bone metabolism assessments.
* Pregnancy or breastfeeding.
* Inability or unwillingness to provide informed consent or to comply with study procedures.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Change in Bone Mineral Density (BMD) | 9 months
  Assessed by DXA (Dual-Energy X-Ray Absorptiometry) scans

SECONDARY OUTCOMES:
Change in Serum Osteocalcin Levels | 9 months
Change in Bone Turnover Markers | 9 months
  Serum C-Terminal Telopeptide (CTX): Measured in ng/mL as a marker of bone resorption.
  Serum Procollagen Type I N-Terminal Propeptide (P1NP): Measured in ng/mL as a marker of bone formation.
  Each marker will be reported separately as the mean change from baseline to 9 months.
Adverse Events and TolerabilityIncidence of Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 9 months
  The number and percentage of participants experiencing treatment-related adverse events will be recorded over the 9-month period. Adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Change in Serum 25(OH) Vitamin D Levels | 9 months
Change in Patient-Reported Quality of Life as Measured by the Short Form-36 Health Survey (SF-36) | 9 months
  Patient-reported quality of life will be assessed using the Short Form-36 Health Survey (SF-36), which generates two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each score ranges from 0 to 100, with higher scores indicating a better quality of life. The outcomes will be reported as the mean change in the PCS and MCS scores from baseline to 9 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Center For New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No